CLINICAL TRIAL: NCT01454687
Title: Grafting of Epidermolysis Bullosa Wounds Using Cultured Revertant Autologous Keratinocytes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alfred Lane, Professor, Departments of Dermatology and Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 22005
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Grafting of Autologous Cultured Revertant Keratinocytes — Grafting of two to four epidermal sheets 40cm2 - 50cm2 onto wounded areas

SUMMARY:
The term epidermolysis bullosa (EB) is used to describe a group of genetic skin diseases associated with skin weakness, blisters, and chronic wounds. "Revertant mosaicism" means that there are two genetically different populations of cells due to spontaneous mutations. Some EB patients have normal, non-fragile skin patches which may be areas of revertant mosaicism. In the revertant areas, the proteins function normally, like non-EB skin. In this study, we plan to culture cells from the revertant areas and graft them on to the wounded areas.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of EB (simplex, junctional or dystrophic)
* Areas of revertant skin that has been confirmed by biopsy
* 18 years or older subject willing and able to give consent
* Confirmation of EB diagnosis by immunofluorescence (IF), electron microscopy (EM), and genetic testing confirming mutation
* At least 100 to 200 cm2 of open erosions on the trunk and/or extremities suitable for skin grafting
* Able to undergo adequate anesthesia to allow grafting procedures to take place

Exclusion Criteria:

* Medical instability limiting ability to travel to Stanford University Medical Center
* The presence of medical illness expected to complicate participation and/or compromise the safety of this technique
* Active infection with HIV, hepatitis B, or hepatitis C
* Active infection in the area that will undergo grafting
* Evidence of a systemic infection
* Current evidence or a history of skin cancer in the area that will undergo grafting
* Active drug or alcohol addiction
* Hypersensitivity to vancomycin or amikacin
* Receipt of chemical or biological study product for the specific treatment ofEB in the past six months
* Positive pregnancy test or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Expression of the correct protein at the basement membrane zone | Week 52
Engraftment and healing of wounds with genetically revertant keratinocytes | Week 52

SECONDARY OUTCOMES:
Engraftment and healing of wounds with genetically revertant keratinocytes | Week 8-12
Engraftment and healing of wounds with genetically revertant keratinocytes | Week 25
Expression of correct protein at the basement membrane zone | Week 8-12
Expression of the correct protein at the basement membrane zone | Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Lane, MD, Principal Investigator — Stanford University